CLINICAL TRIAL: NCT01533597
Title: Comparison of the Efficacy of Solifenacin With or Without Tamsulosin in Adult Women With OAB: A Prospective Randomized Multicenter Study
Brief Title: The Efficacy of Solifenacin With or Without Tamsulosin in Adult Women With Overactive Bladder (OAB)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Kwang-Woo Lee, MD, Clinical Professor, Soonchunhyang University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bomnal study
Record Dates: First submitted 2012-02-02; First posted 2012-02-15 (Estimated); Results first posted 2015-01-27 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Overactive Bladder
Keywords: Overactive bladder; Solifenacin succinate; Tamsulosin
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate; Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Solifenacin (Active Comparator)
  Interventions: Drug: Solifenacin
- Solifenacin plus Tamsulosin (Experimental)
  Interventions: Drug: Solifenacin plus Tamsulosin

INTERVENTIONS:
Drug: Solifenacin — Solifenacin (5mg, qd, oral)
  Other Names: Vesicare
  Arms: Solifenacin
Drug: Solifenacin plus Tamsulosin — Solifenacin (5mg, qd, oral) plus Tamsulosin (0.2mg, qd, oral)
  Other Names: Vesicare; Harnal
  Arms: Solifenacin plus Tamsulosin

SUMMARY:
The aim of the study is to investigate if the combination therapy consisting of anticholinergics plus alpha-blockers could be beneficial for women suffering from Overactive Bladder (OAB).

DETAILED DESCRIPTION:
Overactive bladder (OAB) describes the symptom complex of urgency, with or without urge incontinence, usually with frequency and nocturia.

The lower urinary tract is innervated by both the parasympathetic and the sympathetic nervous system, that act via muscarinic and adrenergic receptors, respectively.

Antimuscarinics are mainly used for the treatment of patients with OAB, especially women. Other than antimuscarinics, a1-blockers have been shown in several clinical reports to be useful in treating DO caused by neurological diseases.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 20 ≤ and < 70 years
* History of OAB symptoms for ≥ 3 months
* International Prostate Symptom Score (IPSS) ≥ 8 points at Screening and more than 3 in total score and 2 in Q 3 index from OABSS questionnaire
* An average of ≥ 8 micturitions per 24 hours and ≥ 1 urgency (defined as a level of 3 to 5 in a 5 point Urinary Sensation Scale) episode (with or without incontinence) per 24 hours as documented in a 3-day micturition diary

Exclusion Criteria:

* Uroflowmetry - Q max ≤ 10 mL/sec, or Post Void Residual Volume ≥ 15% of voided urine
* Any condition that would contraindicate their usage of anticholinergics or alpha blockers
* History of lower urinary tract surgery (e.g. incontinence surgery or electrostimulation)
* History of stress urinary incontinence or urinary retention
* History of interstitial cystitis, bladder outlet obstruction or other significant genitourinary disorder
* Pregnant or nursing women
* Current urinary tract infection
* Neurological bladder dysfunction
* Treatment with drugs that may interfere with CYP3A4 metabolic function
* Significant hepatic or renal disease
* Any other condition which, in the opinion of the investigator, makes the patient unsuitable for inclusion

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kwang Woo Lee, Ph.D, Principal Investigator — Soonchunhyang University Hospital
Locations (1):
- Soonchunhyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do, South Korea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Solifenacin | Solifenacin Plus Tamsulosin
Started | 35 | 35
Completed | 29 | 25
Not Completed | 6 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Solifenacin | Solifenacin Plus Tamsulosin | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 34 | 66
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (8.2) | 52.3 (13.8) | 52.2 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 70
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Number of Micturition Episodes Per 24 Hours
Time Frame: at week 24 relative to baseline
Measure: Mean (95% Confidence Interval); unit: episodes
Arm/Group | Solifenacin | Solifenacin Plus Tamsulosin
Number analyzed (Participants) | 29 | 25
episodes | -1.9 [-2.5 to -1.2] | -2.2 [-3.0 to -1.4]

2. Secondary Outcome: Numeric Change of Urgency Episodes Per 24 Hours
Time Frame: at week 24 relative to baseline
Measure: Mean (95% Confidence Interval); unit: episodes
Arm/Group | Solifenacin | Solifenacin Plus Tamsulosin
Number analyzed (Participants) | 29 | 25
episodes | -2.4 [-3.6 to -1.2] | -2.1 [-2.7 to -1.5]

3. Secondary Outcome: Change in Total Score of OABSS
Description: Total Score of OABSS(Overactive Bladder Symptom Score) is the sum of 4 questions, ranging from 0 (best possible outcome) to 15 (worst possible outcome)
Time Frame: at week 24 relative to baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Solifenacin | Solifenacin Plus Tamsulosin
Number analyzed (Participants) | 29 | 25
units on a scale | -3.1 [-4.2 to -2.0] | -3.5 [-4.3 to -2.7]

4. Secondary Outcome: Change in Score of IPSS
Description: Total Score of IPSS(International Prostate Symptom Score) is the sum of 7 questions, ranging from 0 (best possible outcome) to 35 (worst possible outcome). The 7 symptom questions include feeling of incomplete bladder emptying, frequency, intermittency, urgency, weak stream, straining and nocturia, each referring to during the last month, and each involving assignment of a score from 0 to 5 for a total of maximum 35 points.
Time Frame: at week 24 relative to baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Solifenacin | Solifenacin Plus Tamsulosin
Number analyzed (Participants) | 29 | 25
units on a scale | -7.7 [-10.4 to -5.1] | -8.3 [-10.3 to -6.3]

5. Secondary Outcome: Change of PVR
Description: Change from baseline in Post-Void Residual (PVR) volume
Time Frame: at week 24 relative to baseline
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | Solifenacin | Solifenacin Plus Tamsulosin
Number analyzed (Participants) | 29 | 25
mL | 13.2 [8.7 to 17.6] | 10.8 [6.9 to 14.7]

6. Secondary Outcome: Change of Qmax
Description: maximal urinary flow rate (Qmax) assessed by uroflowmetry
Time Frame: at week 24 relative to baseline
Measure: Mean (95% Confidence Interval); unit: mL/sec
Arm/Group | Solifenacin | Solifenacin Plus Tamsulosin
Number analyzed (Participants) | 29 | 25
mL/sec | 1.1 [-0.6 to 2.7] | 2.1 [-0.5 to 4.8]

ADVERSE EVENTS:
Time Frame: 24weeks
Arm/Group | Solifenacin | Solifenacin Plus Tamsulosin
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 2/35 | 2/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Solifenacin (N=35) | Solifenacin Plus Tamsulosin (N=35)
constipation (Gastrointestinal disorders) | 0 | 1
dry mouth (Endocrine disorders) | 2 | 1

LIMITATIONS AND CAVEATS:
small study population

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No